CLINICAL TRIAL: NCT05314556
Title: Effectiveness of Group Psychotherapy in Patients With Narcolepsy Type 1
Brief Title: Group Psychotherapy in Narcolepsy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Nicolas Germann, Principal Investigator, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01324
Record Dates: First submitted 2022-03-15; First posted 2022-04-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Narcolepsy Type 1
Keywords: Narcolepsy Type 1; Narcolepsy; Narcolepsy with cataplexy; Group psychotherapy; Group therapy; Psychotherapy
MeSH Terms: conditions — Narcolepsy | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Group psychotherapy
  Interventions: Behavioral: Group psychotherapy

INTERVENTIONS:
Behavioral: Group psychotherapy — Additional group psychotherapy for patients with narcolepsy type 1 with standard medication

SUMMARY:
The aim of this pilot study is to test the benefit of behavior therapy-oriented, method-integrated psychotherapy in an outpatient group setting in patients with narcolepsy type 1. Therefore we collect and evaluate initial data on its effectiveness on the disease in terms of specific symptomatology, emotion regulation, health-related quality of life, and disease processing/acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed narcolepsy type 1 according to AASM, examined by an experienced sleep physician including history, clinical examination, polysomnographic examination (PSG) with a multiple sleep latency test (MSLT), possibly also including determination of HLA DQB1 * 062 and orexin A / hypocretin 1
* Age between 18 and 65 years
* Signed informed consent
* Exclusion of other clinically relevant organic sleep disorders by means of polysomnography (AHI>10/h)

Exclusion Criteria:

* Presence of severe psychiatric comorbidity
* Other psychotherapy during the study period
* Change of medication used for narcolepsy therapy shortly before the start and during the study period including follow-up measurement. In this case, patients may still complete group therapy, but the data will not be included in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue (Severity) | Week 0-24
  German version of the questionnaire "Fatigue Severity Scale" (FSS; Valko et al., 2008)
Daytime sleepiness | Week 0, Week 6, Week 12, Week 24
  German version of the questionnaire "Epworth Sleepiness Scale" (ESS; Johns, 1991)
Sleep quality | Week 0-24
  German version of the questionnaire "Pittsburgh Sleep Quality Index" (PSQI; Buysse et al., 2008)
Emotion regulation | Week 0-24
  German questionnaire "Fragebogen zur Erhebung der Emotionsregulation bei Erwachsenen" (FEEL-E; Grob et al., 2014)

SECONDARY OUTCOMES:
Disease processing, acceptance & coping | Week 0, Week 6, Week 12, Week 24
  German questionnaire "Freiburger Fragebogen zur Krankheitsverarbeitung" (FKV-LIS-SE; Muthny, 1989)
Anxiety & depression | Week 0, Week 6, Week 12, Week 24
  German version of the questionnaire "Hospital Anxiety and Depression Scale" (HADS; Herrmann et al., 1995; Herrmann-Lingen et al., 2011; Zigmond & Snaith, 1983)
Health-related quality of life (HRQOL) | Week 0-24
  German version of the questionnaire "Short Form 12 Health Survey" (SF-12; Morfeld et al., 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar A Schmid, Dr. med, Principal Investigator — Klinik für Psychosomatik und Konsiliarpsychiatrie, Kantonsspital St.Gallen
Locations (1):
- Clinic for Psychosomatic Medicine, Cantonal Hospital St.Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No